CLINICAL TRIAL: NCT07170085
Title: Positioning of Children With Acute Respiratory Insufficiency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HCA-PC
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Acute Respiratory Disease
Keywords: positioning
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supine-prone (Experimental): first supine position, then prone position
  Interventions: Other: positioning
- prone-supine (Experimental): first prone position, then supine position
  Interventions: Other: positioning

INTERVENTIONS:
Other: positioning — The children will be positioned in the supine and prone position

SUMMARY:
Acute respiratory insufficiency is one of the most common causes of hospitalization and death among young children. It often affects small children who, due to infections with RSV (respiratory syncytial virus), other cold viruses, or bacteria, experience difficulty breathing, rapid breathing, increased heart rate, low oxygen levels in the blood, and reduced appetite. If left untreated, a child can become exhausted, lose consciousness, and ultimately die from the condition. Children with severe acute respiratory insufficiency occupy most of the acute care beds in the pediatric wards of hospitals during the winter months. Some children are treated simply with saline inhalations, nasal saline drops, and suctioning of the nose, but many require respiratory support in the form of Continuous Positive Airway Pressure (CPAP) or high-flow oxygen therapy.

In adults, it has been observed that prone positioning can improve blood oxygenation compared to supine positioning in cases of acute respiratory insufficiency.

The purpose of this study is to investigate whether there are benefits or drawbacks to positioning small children admitted for difficulty breathing due to respiratory infections in a prone position instead of a supine position.

The study will include a total of 40 children with acute airway disease who have been prescribed respiratory support in the form of CPAP or high-flow oxygen. The study will last a total of 2 hours and will not involve any uncomfortable procedures or pose any risks to the child.

The Study Itself:

Once the child has CPAP or high-flow oxygen administered via the nose, the child will be positioned for 1 hour in the prone position and 1 hour in the supine position. The order will be random and determined by lottery. A nurse will record the child's breathing in both the prone and supine positions. After the two hours, the child will be placed in the supine position, which is standard practice in the department. The child will have a pulse oximeter on both during the study and afterwards.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether there are benefits or drawbacks to positioning small children admitted for difficulty breathing due to respiratory infections in a prone position instead of a supine position.

Hypothesis:

Children under 1 year of age with acute respiratory insufficiency undergoing CPAP or High-Flow oxygen therapy will have improved respiratory function when positioned in the prone position compared to the supine position, as assessed by respiratory rate and symptom score.

The study will include a total of 40 children with acute airway disease who have been prescribed respiratory support in the form of CPAP or high-flow oxygen.

. Method: The study is designed as an open-label, randomized crossover study. The intervention involves positioning: 1 hour in the prone position and 1 hour in the supine position while the child receives treatment with CPAP or High-Flow oxygen.

The study will enroll children hospitalized with infection-triggered acute respiratory insufficiency, who, based on a clinical physician's assessment, are indicated for treatment with either CPAP or High-Flow oxygen. They will be randomized to either prone positioning followed by supine positioning or supine positioning followed by prone positioning upon initiation of respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-12 months
* Clinical respiratory infection
* Physician-ordered High-Flow oxygen or CPAP
* Consent from the legal guardian

Exclusion Criteria:

* Significant chronic pulmonary, cardiac, or neurological disorders
* Children admitted to intensive care

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
m-WCAS | one hour
  Modified Wood's Clinical Asthma Score (mWCAS) a combined score of saturation, inspiratory wheezes, expiratory wheezes, retractions, general condition, each scored 1-4, with 1 being the best and 4 being the worst
respiratory rate | 1 hour
  respiration per minute

SECONDARY OUTCOMES:
saturation | 1 hour
  percent
pulse | 1 hour
  hearth rate
apneas | 1 hour
  Number of apneas >10 seconds

CONTACTS AND LOCATIONS:
Overall Officials: The Research Unit Hans Christian Andersn Children´s Hospital, Study Chair — Odense University Hospital
Locations (1):
- Hans Christian Andersen´s Childrens Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No